CLINICAL TRIAL: NCT04600362
Title: An Investigator-initiated, Multi-center, Randomized, Double-blind, Placebo Controlled Study of Dupilumab to Demonstrate Efficacy in Subjects With Nummular Eczema
Brief Title: Study of Dupilumab to Demonstrate Efficacy in Subjects With Nummular Eczema
Acronym: DUPINUM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: University Hospital Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGZ-2018-12012
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-06

CONDITIONS: Nummular Eczema
Keywords: Nummular Eczema; Dermatitis; Skin Diseases; Dupilumab; Anti-Inflammatory-Sgents
MeSH Terms: conditions — Dermatitis; Skin Diseases | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: This is an investigator-initiated, multi-center, prospective, randomized, double-blind, interventional phase II study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dupilumab (Experimental): Patients randomized to this arm will receive two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by single 300 mg injection of Dupilumab every 2 weeks (q2w) from week 2 to week 16.
  Interventions: Drug: Experimental: Dupilumab 300 MG/2 ML Subcutaneous Solution [DUPIXENT]
- Placebo (Placebo Comparator): Patients randomized to this arm will receive identically matching doses of placebo. Two subcutaneous injections of placebo as a loading dose (to mimic the experimental Dupilumab arm) on Day 1 followed by a single injection q2w from Week 2 to Week 16.
  Interventions: Drug: Experimental: Dupilumab 300 MG/2 ML Subcutaneous Solution [DUPIXENT]

INTERVENTIONS:
Drug: Experimental: Dupilumab 300 MG/2 ML Subcutaneous Solution [DUPIXENT] — Subcutaneous

SUMMARY:
Nummular eczema (NE) is an idiopathic chronic inflammatory skin disease that occurs throughout all life periods. Diagnosis is made primarily clinically in correlation with histological findings. Treatment of NE is difficult. Standard treatment consists of the use of emollients, topical as well as systemic corticosteroids and phototherapy. Nevertheless, remission is hard to achieve and relapse occurs often. Patients usually suffer from severe pruritus and reduced quality of life. Therefore, new therapeutic strategies are urgently needed.

Dupilumab (Dupixent®), a monoclonal antibody inhibiting the IL-4 and IL-13 pathway by targeting the IL-4-receptor, has been approved for the treatment of moderate-to-severe atopic dermatitis (AD). Since there is an overlap between AD and NE with both being caused by impaired epidermal barrier, broad immune-mediated inflammation and microbial skin colonization, using Dupilumab in NE seems to be promising.

DETAILED DESCRIPTION:
This study aims on investigating the efficacy of Dupilumab in NE patients. The primary endpoint is the percent change in Eczema Area and Severity Index (EASI) score from baseline to week 16.

Secondary endpoints include the number of patients achieving an improvement (decrease) in Physician Global Assessment (PGA) by two or more points at week 16 as compared to week 0 or achieving an absolute PGA of 0 or 1 at Week 16, the EASI 50 score at week 16, the change from baseline in transepidermal waterloss (TEWL) at week 16, significant histological improvement at week 16, change from baseline in the reduction of the use of topical steroids at week 16, change form baseline in the Dermatology Life Quality Index (DLQI) at week 16, change from baseline in Pruritus Visual Analog Scale (VAS), change from baseline in the global satisfaction subscale of the treatment satisfaction questionnaire for medication (TSQM) score at week 16 and the safety of Dupilumab.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically confirmed diagnosis of NE.
2. Biopsy-proven, meaning histology consistent with eczema (including PAS-staining).
3. EASI score ≥ 10.
4. PGA ≥ 3 on a 5 point scale.
5. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
6. Female participants who are not capable of bearing children or who use a method of contraception that is medically approved by the health authority of the respective country at screening. Effective contraception (CTFG guideline) for women of childbearing potential should be used throughout the study, including during the follow-up period or at least 120 days after last dose, whichever is longer (elapse of 4-5 half-lives). The event of pregnancy, Dupilumab should be immediately discontinued.
7. History of continuous use of at least mid-potency topical steroids for the last 8 weeks.
8. Age 18-85 years of age, body weight ≥ 40 kg and ≤ 160 kg.
9. Signed informed consent from patient.

Exclusion Criteria:

1. Permanent severe diseases, especially those affecting the immune system.
2. Pregnancy or breast feeding.
3. Active chronic or acute infection requiring systemic treatment within 2 weeks before the baseline visit, independent from of the cuntaneous dysbiosis found in NE.
4. Treatment with an investigational drug within 8 weeks before the baseline visit.
5. Treatment with a live (attenuated) vaccine within 12 weeks before the baseline visit.
6. Diagnosed active endoparasitic infections or at high risk of these infections.
7. Evidence of severe renal dysfunction 8.Evidence of significant hepatic disease 9.Patients who are considered potentially unreliable or where it is envisaged the patient may not consistently attend scheduled study visits. 10.Inability or unwillingness to undergo repeated venipuncture (e.g., because of poor tolerability or lack of access to veins).

11.Inability or unwillingness to undergo repeated punch biopsies. 12.History of allergy to any component of the study medication. 13.Evidence of acute contact dermatitis at screening. 14.Evidence of Zink deficiency defined as Zink level < 20 µg/dL in serum. 15.History of important side effects of medium potency topical corticosteroids (eg, intolerance to treatment, hypersensitivity reactions*, significant skin atrophy, systemic effects), as assessed by the investigator or patient's treating physician.

16. ≥30% of the total lesional surface located on areas of thin skin that cannot be safely treated with medium potency TCS (eg, face, neck, intertriginous areas, genital areas, areas of skin atrophy) at baseline.

17. Planned or anticipated use of any prohibited medications and procedures during study treatment.

18. Known history of human immunodeficiency virus (HIV) infection. 19. Established diagnosis of Hepatitis B viral infection at the time of screening.

20. Established diagnosis of hepatitis C viral infection at the time of screening.

21. History of past or current tuberculosis or other mycobacterial infection. 22. Presence of skin comorbidities that may interfere with study assessments. 23. Malignancy within 5 years of the screening visit excluding local cutaneous squamous cell 24. Severe concomitant illness(es) 25. Any other medical or psychological condition including relevant laboratory abnormalities at Screening 26. Planned major surgical procedure during the patient's participation in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
EASI | From baseline to week 16.
  The primary endpoint is the percent change in Eczema Area and Severity Index (EASI) score.

SECONDARY OUTCOMES:
PGA | at week 16 as compared to week 0
  Number of Patients Achieving an Improvement (Decrease) in Physician Global Assessment (PGA) by two or more points
PGA | at Week 16.
  Number of Patients achieving an absolute PGA of 0 or 1
EASI | From baseline to week 16
  The proportion of subjects who achieve at least a 50% reduction in the EASI score
TEWL | From baseline to week 16
  Restoration of epidermal barrier function assessed by TEWL (Transepidermal Waterloss) will be measured using AquaFlux BIOX.
histological improvement | From baseline to week 16
  Assessed by reduction of epidermal thickness > 30% or reduction of inflammatory infiltrate > 50 %
Reduction of the Use of Topical Steroids | From baseline to week 16
  Prior to randomization and during the treatment, average application rate of class II topical steroids (standard medication "prednicarbate") per day will be calculated
DLQI | Total Score at Week 16
  Change from Baseline in the Dermatology Life Quality Index (DLQI)
VAS | Total Score at Week 16
  Pruritus Visual Analog Scale
TSQM | Total Score at Week 16
  Global Satisfaction Subscale of the Treatment Satisfaction Questionnaire for Medication
Adverse Events | From baseline to week 16
  Type, incidence, severity, and relationship of the AEs to study medication

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Biedermann, Prof.Dr.med., Principal Investigator — Klinikum re. Isar, Technische Universität München, Dermatologie
Locations (1):
- Klinikum re. Isar Dermatology, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
All participant data collected during the clinical trial (pseudonymized)
Supporting Information: CSR
Time Frame: A year later according to LPLV
Access Criteria: Publikation

REFERENCES:
- [Derived] Bohner A, Jargosch M, Muller NS, Garzorz-Stark N, Pilz C, Lauffer F, Wang R, Roenneberg S, Zink A, Thomas J, Theis FJ, Biedermann T, Eyerich S, Eyerich K. The neglected twin: Nummular eczema is a variant of atopic dermatitis with codominant TH2/TH17 immune response. J Allergy Clin Immunol. 2023 Aug;152(2):408-419. doi: 10.1016/j.jaci.2023.04.009. Epub 2023 Apr 27. PMID 37119871